CLINICAL TRIAL: NCT01532115
Title: A Randomized, Double-blind, Placebo-controlled and Open-label Active-controlled, 4-period Crossover Trial to Evaluate the Effect of BIA 9-1067 on Cardiac Repolarization in Healthy Adult Men and Women
Brief Title: Effect of BIA 9-1067 on Cardiac Repolarization in Healthy Adult Men and Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BIA-91067-111
Record Dates: First submitted 2012-01-23; First posted 2012-02-14 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; BIA 9-1067
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- BIA 9-1067 (Experimental)
  Interventions: Drug: BIA 9-1067
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- moxifloxacin (Active Comparator)
  Interventions: Drug: moxifloxacin

INTERVENTIONS:
Drug: BIA 9-1067 — 50 mg and 800 mg of BIA 9-1067 (single-dose)
  Arms: BIA 9-1067
Drug: Placebo — single-dose
  Arms: Placebo
Drug: moxifloxacin — 400 mg moxifloxacin (single-dose)
  Arms: moxifloxacin

SUMMARY:
The purpose of this study is to evaluate the effect of BIA 9-1067 on the cardiac repolarization in adult healthy men and women volunteers.

DETAILED DESCRIPTION:
Single-centre, randomized, double-blind, placebo-controlled and open-label active-controlled, 4-period crossover trial in healthy male and female subjects

ELIGIBILITY:
Inclusion Criteria:

* A signed and dated informed consent form before any study-specific screening procedure was performed,
* Healthy male or female 18 to 55 years of age. Women had to be postmenopausal (more than 12 months since last period); surgically sterile (hysterectomy or tubal ligation or bilateral oophorectomy at least 6 months prior to enrollment); using an intrauterine device; a non-hormonal double barrier contraceptive method (i.e., diaphragm or spermicide plus male condom) for the duration of the trial and with a negative pregnancy test at screening and upon each check-in to the study facility,
* Had a BMI within the range of 18-30 kg/m2,
* Able to communicate effectively with the study personnel,
* Had no significant disease or abnormal laboratory values as determined by medical history, physical examination or laboratory evaluations, conducted at the screening visit and on admission to the clinic,
* Had a normal 12-lead electrocardiogram, without any clinically significant abnormalities of rate, rhythm or conduction,
* Non-smokers or ex-smokers for at least 3 months,
* Adequately informed of the nature and risks of the study and gave written informed consent prior to study entry.

Exclusion Criteria:

* Known hypersensitivity or allergy to moxifloxacin, BIA 9-1067 or related compounds such as tolcapone or entacapone,
* Women who were pregnant or breastfeeding,
* Any disease or condition (medical or surgical) which, in the opinion of the Investigator, might have compromised the hematologic, cardiovascular, pulmonary, renal, gastrointestinal, hepatic, or central nervous system; or other conditions that might have interfered with the absorption, distribution, metabolism or excretion of study drug, or would have placed the subject at increased risk,
* A sustained supine systolic blood pressure > 140 mmHg or < 100 mmHg or a diastolic blood pressure > 95 mmHg at screening or baseline,
* A resting ECG heart rate of < 50 bpm or > 100 bpm,
* An abnormal screening ECG indicating a second- or third-degree AV block, or one or more of the following: QRS > 110 milliseconds (ms), QTc (Fridericia correction) > 450 ms for male and 470 ms for females, PR interval > 240 ms. Any rhythm other than sinus rhythm, which was interpreted by the Investigator to be clinically significant,
* The presence of abnormal laboratory values which were considered clinically significant by the Investigator,
* Positive screen for Hepatitis B (HbsAg, Hepatitis B Surface Antigen), Hepatitis C (anti HCV, Hepatitis C Antibody), or HIV (anti-HIV 1/2),
* Received an investigational drug within a period of 30 days prior to enrolment in the study,
* Received any drug therapy, excluding hormonal contraceptives, within 2 weeks prior to administration of the first dose of any study-related treatment. This exclusion was extended to 4 weeks for any drugs known to induce or inhibit hepatic drug metabolism,
* Consumption of alcohol within 48 hours prior to dose administration or during any inpatient period,
* A positive urine drug screen including or a positive alcohol breath test,
* Any history of alcohol abuse, illicit drug use, significant mental illness, physical dependence to any opioid, or any history of drug abuse or addiction,
* A history of difficulty with donating blood,
* Donated blood or blood products within 45 days prior to enrollment,
* History of tendonitis or tendon rupture associated with treatment with quinolone antibiotics,
* Subjects with, or with a history of, additional risk factors for Torsades de Pointes (e.g., heart failure, hypokalemia), or a family history of long QT syndrome or family history of sudden death.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2010-05; Primary Completion 2010-10 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Number and percentage of subjects with ECG abnormalities | 56 days
  Through standard 12-lead ECGs assess the effect BIA 9-1067 on heart rate(HR),These ECGs were centrally reviewed. Cardiac effects were assessed through an evaluation of QT, QTc (QTcI, QTcB, and QTcF), PR, QRS interval duration, HR, and morphological changes.

SECONDARY OUTCOMES:
Number of participants with Adverse Events | 56 days
  assessment of safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Claude Homery, MD, Principal Investigator — Biotrial
Locations (1):
- Biotrial, 7-9 rue Jean-Louis Bertrand, Rennes, France